CLINICAL TRIAL: NCT01648179
Title: A Single Dose, Open Label, Randomized, Balanced, Crossover Study to Assess the Relative Bioavailability of ThreeFormulations and Food Effect on GSK1322322 in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Three Formulations and Food Effect on GSK1322322 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116595
Record Dates: First submitted 2012-06-07; First posted 2012-07-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Infections, Bacterial
Keywords: GSK1322322, relative bioavailability, healthy subjects, open label, food effect, weight effect
MeSH Terms: conditions — Bacterial Infections | interventions — GSK1322322; Powders; Injections; Tablets; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK1322322 IV formulation (Experimental): Subjects will be randomized in a cross over fashion to receive the GSK1322322 administered via IV formulation
  Interventions: Drug: GSK1322322 (mesylate salt) Powder for Injection
- GSK1322322 Wet milled Tablet (Fasted) (Experimental): Subjects will be randomized in a cross over fashion to receive the GSK1322322 administered via Wet milled Tablet (Fasted)
  Interventions: Drug: GSK1322322 (freebase) tablets
- GSK1322322 Oral mesylate salt solution (Experimental): Subjects will be randomized in a cross over fashion to receive the GSK1322322 administered via Oral mesylate salt solution
  Interventions: Drug: GSK1322322 (mesylate salt) Powder for Oral Solution
- GSK1322322 Wet milled Tablet (Fed) (Experimental): Subjects will be randomized in a cross over fashion to receive the GSK1322322 administered via Wet milled Tablet (Fed)
  Interventions: Drug: GSK1322322 (freebase) tablets FED

INTERVENTIONS:
Drug: GSK1322322 (mesylate salt) Powder for Injection — 1500 mg (mesylate salt) as free base, dissolved in sterile water for injection to a concentration of 100 mg/mL free base equivalent and sterilized via filtration. 15 mL of solution, equivalent to 1500 mg GSK 1322322, is the diluted into 0.9% Sodium Chloride Injection prior to infusion
  Arms: GSK1322322 IV formulation
Drug: GSK1322322 (freebase) tablets — 500 mg tablets for a 1500 mg total single dose (3 tablets). Taken with 240 mL of water
  Arms: GSK1322322 Wet milled Tablet (Fasted)
Drug: GSK1322322 (mesylate salt) Powder for Oral Solution — 1500 mg as a free base, dissolved in purified water to a concentration of 100 mg/mL free base equivalent. 15 mL of solution, equivalent to1500 mg GSK1322322 is administered orally with 225 mL of water
  Arms: GSK1322322 Oral mesylate salt solution
Drug: GSK1322322 (freebase) tablets FED — Drug 500 mg tablets for a 1500 mg total single dose (3 tablets) (FED moderate fat meal) Taken with 240 mL of water
  Arms: GSK1322322 Wet milled Tablet (Fed)

SUMMARY:
This study is an open-label, randomized, single dose, four period, balanced crossover study to assess in eligible healthy male or female subjects.

DETAILED DESCRIPTION:
This study is an open-label, randomized, single dose, four period, balanced crossover study to assess in eligible healthy male or female subjects:

* The relative bioavailability of the wet milled GSK1322322 tablet formulation with and without food compared to an oral mesylate salt solution.
* The effect of body weight on the pharmacokinetics of GSK1322322 when given either orally or IV.
* The absolute bioavailability of the wet milled tablet and the oral mesylate salt solution compared to the IV formulation.

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTcB < 450 msec; or QTcB < 480 msec in subjects with Bundle Branch Block.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female (of non childbearing potential) between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample withsimultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory].
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the final follow up visit.
* Body weight ≥ 40 kg (Refer to Table 3 for weight stratification details).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety due to potential drug interaction.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.10. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive [serum or urine] hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Males Females Heart rate <45 and >100 bpm <50 and >100 bpm PR Interval <120 and >220 msec QRS duration <70 and >120 msec QTc interval (Bazett) >450 msec

  * Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).
  * Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (≥3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To estimate the relative bioavailability of wet milled tablet formulations of GSK1322322 with and without food as compared to an oral mesylate salt solution following single doses in healthy subjects. | 72 Hours
  GSK1322322 AUC(0-∞) and Cmax following wet milled tablet formulation administered with and without moderate fat/calorie meal. GSK1322322 AUC(0-∞) and Cmax following oral mesylate salt solution administration.
To estimate the effect of body weight on the pharmacokinetics of GSK1322322 formulations (IV and oral) following single dose administration to healthy subjects. | 72 Hours
  GSK1322322 AUC(0-∞) and Cmax in each body weight group following IV or oral formulation administration to assess effect of body weight.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of GSK1322322 after single doses of each formulation in healthy subjects. | 14 Days
  Safety parameters including adverse events, clinical laboratory tests, concomitant medications, electrocardiograms, and vital signs.
To estimate the absolute bioavailability of the different oral formulations of GSK1322322 as compared to IV mesylate salt formulation following single doses in healthy subjects. | 72 Hours
  GSK1322322 AUC(0-∞) following different oral formulations (oral mesylate salt solution and wet milled tablet) versus IV formulation to assess absolute bioavailability. GSK1322322 pharmacokinetic parameters will be computed with noncompartmental analysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study116595 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116595?search=study&#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116595 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register